CLINICAL TRIAL: NCT03705702
Title: Effects of Behavioral Intervention to Increase Physical Activity on the Asthma Clinical Control: a Randomized Controlled Trial
Brief Title: Behavioral Intervention to Increase Physical Activity in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIPAA; 2016/17093-0 (Other Grant/Funding Number: São Paulo Research Foundation (FAPESP))
Record Dates: First submitted 2018-10-04; First posted 2018-10-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Physical activity; Behavioral intervention; Asthma clinical control
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Early Intervention, Educational; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All the measurements will be performed by a blinded professional, who will be masked from randomization and other results. For each test, the same investigator will be maintained before and after the intervention. The participants will know what treatment they will receive, but they don't will know what intervention belongs to the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Active Comparator): The intervention of active comparator will be education program plus behavioral intervention through physical activity counseling program combined with a monitoring-and-feedback tool.
  Interventions: Other: Education Program; Behavioral: Behavioral intervention
- Control Group (CG) (Sham Comparator): The intervention of sham comparator will be an education program in asthma and physical activity recommendations.
  Interventions: Other: Education Program

INTERVENTIONS:
Other: Education Program — The educational program will consist of 2 classes held once a week, each lasting 90 minutes. The classes will be based on an education videotape, presentations and group discussions. The first class will address the asthma education, which will include information about the pathophysiology of asthma, medication and peak flow meter instructions, self-monitoring techniques, environmental control techniques and avoidance strategies. The second class will be about the current international physical activity recommendations and the importance and benefits of being physically active and maintain a healthy lifestyle.
Behavioral: Behavioral intervention — The behavioural intervention will be performed in 8 weekly goal-setting consultation, face-to-face, each lasting 40 minutes. Patients will be offered a commercially-available activity tracker to wear during 3 days prior to each consultation. According to their own PA data and the behavioural change stage, an individual action plan will be established with realistic goals to increase PA. Each participant will receive individual counselling with the goal of increasing participation in PA and reducing their sedentary time. Techniques such as weekly goal-setting, motivational interviewing, activity tracker vibration instructions, self-management, positive reinforcement, relapse prevention and strategies to overcome barriers will be included.
  Arms: Intervention Group (IG)

SUMMARY:
The health benefits of physical activity (PA) are well documented and include improving in cardiovascular, obesity, mental health and all-cause mortality. Although higher levels of activity in patients with asthma are also associated with better outcomes, patients still avoid physical activity due to concern about exacerbating their asthma symptoms by the exercise induced bronchoconstriction (EIB), sustaining a vicious cycle of inactivity and worse asthma control. Many studies have reported the benefits of supervised exercise training on several asthma outcomes, such as exacerbations, asthma control, cardiopulmonary fitness, airway inflammation and psychosocial symptoms; however, the translation of the improvements in the exercise capacity into increments in PA levels is less evident and still controversial. Therefore, the hypothesis of this study is that behavioural interventions using strategies based on well-established psychosocial models are effective in increasing physical activity levels and decrease sedentary behaviour in adults with asthma, which will be associated with improvements in the asthma control.

DETAILED DESCRIPTION:
This is prospective and randomized controlled trial (RCT) with 2 arms and blinded outcome assessments. Forty-six moderate or severe patients with asthma under optimized medication will be randomly assigned (computer-generated) into either Control Group (CG) or Intervention Group (IG). Both groups will receive similar educational program. However, only the IG will be submitted to the behavioral intervention through physical activity counseling program combined with a monitoring-and-feedback tool aiming to increase physical activity levels (total of 8 weekly goal-setting consultation, face-to-face, each lasting 40 minutes). Before and after the interventions, clinical control of asthma, physical activity levels, health-related quality of life, asthma exacerbation, levels of anxiety and depression symptoms and anthropometric indices will be assessed. Data about onset of asthma, comorbidities, lung function and asthma medication will be collected from the patient's medical record. The data normality will be analyzed by Kolmogorov-Smirnov, and a two-way ANOVA with repeated measures with appropriate post hoc of Holm-sidak will be used to compare inter and intra-groups differences. The significance level will be set to 5% for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe with diagnosed according to the Global Initiative for Asthma (GINA) 2018
* Poorly controlled asthma (ACQ score > 1.5)
* Sedentary (< 150 min of moderate to vigorous physical activity/week)
* Medical treatment, for at least 6 months
* Clinically stable (i.e., no exacerbation or changes in medication for at least 30 days)

Exclusion Criteria:

* Cardiovascular, musculoskeletal or other chronic lung diseases
* Active Cancer
* Pregnant
* Uncontrolled hypertension or diabetes
* Current smoker or ex smoker (>10 pack-years)
* Psychiatric disease or cognitive deficit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in asthma clinical control | Change from baseline asthma clinical control at 8 weeks of intervention
  Clinical control will be evaluated by the Asthma Control Questionnaire (ACQ). The ACQ contains 7 items rated on a 7-point scale (0 = without limitation, 6 = maximum limitation), with a higher score indicating worse control. Scores lower than 0.75 are associated with good asthma control, whereas scores greater than 1.5 are indicative of poorly controlled asthma, and a change of at least 0.5 points in the ACQ score is regarded as clinically significant.

SECONDARY OUTCOMES:
Change in physical activity levels | Change from baseline physical activity levels at 8 weeks of intervention
  Physical activity and sedentary behaviour will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive days on the hip using an elastic belt. Sedentary behaviour will be quantify by the time spent sedentary (< 100 counts/min).
Change in health related quality of life | Change from baseline health related quality of life at 8 weeks of intervention
  Health related quality of life will be assessed by Asthma Quality Life Questionnaire (AQLQ). The AQLQ consists of 32 items rated on a 7-point scale (1 = great deal, 7 = not at all) divided into the following 4 domains: activity limitations, symptoms, emotional function and environmental stimuli. Higher AQLQ scores indicate a better quality of life, and treatments resulting in a 0.5-point increase in scores following an intervention are considered to be clinically effective.
Change in asthma exacerbation | Change from baseline asthma exacerbation at 8 weeks of intervention
  Asthma exacerbation will be assessed by the following criteria: the use of ≥4 puffs of rescue medication per 24 hours during a 48-hour period, a need for systemic corticosteroids, an unscheduled medical appointment, and either a visit to an emergency room or hospitalization
Change in sleep quality | Change from baseline sleep quality at 8 weeks of intervention
  Sleep quality will be objectively quantified using a movement sensor (ActiGraph, Pensacola, USA) for 7 consecutive nights on the wrist (non-dominant side).

OTHER OUTCOMES:
Pulmonary function | At baseline
  Lung volumes will be assessed by spirometry
Change in anthropometric indexes | Change from baseline anthropometric indexes at 8 weeks of intervention
  Height (m) and weight (kg) will be combined to report BMI (kg/m^2)
Change in body composition | Change from baseline body composition at 8 weeks of intervention
  Waist circumference (cm) and hip circumference (cm) will be combined to report wait to hip ratio (WHR)
Change in psychosocial symptoms | Change from baseline psychosocial symptoms at 8 weeks of intervention
  Symptoms of anxiety and depression symptoms will be assessed by the Hospital Anxiety and Depression scale (HADs), which consists of 14 items divided into 2 subscales (7 for anxiety and 7 for depression). Each item is scored from 0 to 3, with a maximum score of 21 points for each subscale. A score greater than 8/9 in each subscale suggests a diagnosis of either anxiety and/or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of Sao Paulo General Hospital
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Passos NF, Freitas PD, Carvalho-Pinto RM, Cukier A, Carvalho CRF. Increased physical activity reduces sleep disturbances in asthma: A randomized controlled trial. Respirology. 2023 Jan;28(1):20-28. doi: 10.1111/resp.14359. Epub 2022 Sep 6. PMID 36068181
- [Derived] Freitas PD, Passos NFP, Carvalho-Pinto RM, Martins MA, Cavalheri V, Hill K, Stelmach R, Carvalho CRF. A Behavior Change Intervention Aimed at Increasing Physical Activity Improves Clinical Control in Adults With Asthma: A Randomized Controlled Trial. Chest. 2021 Jan;159(1):46-57. doi: 10.1016/j.chest.2020.08.2113. Epub 2020 Sep 12. PMID 32931821